CLINICAL TRIAL: NCT04568109
Title: Effect of Cognitive-behavior Therapy on Panic Symptomatology and the Activation of the Brain's Fear Network to Panic-related Body Symptoms in Patients With Panic Disorder
Brief Title: Effect of Cognitive-behavior Therapy on Fear Responses to Body Symptoms in Patients With Panic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Christane Pané-Farré, Prof. Dr. Christiane Pané-Farré, Philipps University Marburg
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PA_CBT_HV
Record Dates: First submitted 2020-09-17; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Panic Disorder With Agoraphobia; Panic Disorder Without Agoraphobia
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure-based cognitive-behavior therapy (Experimental): Patients are treated in accordance with a manualized protocol (Gloster et al., 2011)
  Interventions: Behavioral: Cognitive-behavior therapy
- Wait-List control condition (No Intervention): Patients are assessed prior to and after a 12-week waiting period. Patients are treated after this 12-week delay.

INTERVENTIONS:
Behavioral: Cognitive-behavior therapy — The manualized protocol (Gloster et al., 2011) comprise of 12 weekly sessions of CBT focusing on therapist-guided interoceptive and in-situ exposure exercises.
  Arms: Exposure-based cognitive-behavior therapy

SUMMARY:
The present study aims to investigate a potential mechanism of successful CBT for panic disorder, i.e., the reduction of excessive anxious apprehension and fear responses to panic-related body symptoms in the context of CBT treatment. In the present non-randomized interventional study, effects of cognitive behavior therapy on reported symptoms and fear responses to panic-related body symptoms are investigated. It is expected that symptom improvement during CBT is associated with a decrease in the activation of the brain's fear network to panic-related body symptoms.

DETAILED DESCRIPTION:
Changes in fear responses to body symptoms in the course of CBT are investigated in patients with PD by applying a highly standardized hyperventilation task (provoking panic-related body symptoms) prior to and after a manualized CBT or a waiting period. Activation of the brain's fear network (defensive activation) is indexed by the potentiation of the startle eyeblink response.

ELIGIBILITY:
Inclusion Criteria:

* current primary diagnosis of panic disorder (with or without agoraphobia) as defined by the criteria of the diagnostic and statistical manual, fourth revision/text revision (DSM-IV-TR) (determined using the Composite International Diagnostic Interview and verified by a certified psychotherapist)
* age 18 - 65 years

Exclusion Criteria:

* current suicidal intent
* any psychotic or bipolar disorder
* borderline personality disorder
* a medical condition that could explain patients' symptoms
* physical contradictions regarding application of exposure-based CBT (e.g., neurological disease)
* Patients has to be on a stable psychopharmacological medication schedule prior to study entry for at least 12 weeks
* Intake of benzodiazepines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2014-04-10 (Actual); Study Completion 2014-05-31 (Actual)

PRIMARY OUTCOMES:
Change in defensive activation to interoceptive threat | change from pre-intervention/pre-waiting period (baseline) to immediately after CBT or waiting period
  Defensive activation to interoceptive threat (induced via a standardized hyperventilation task) is assessed using the startle eyeblink response (measured via electromyographic activity over the left musculus orbicularis oculi) to an acoustic startle probe.
Change in panic symptomatology and severity (PAS) | change from pre-intervention/pre-waiting period (baseline) to immediately after CBT or waiting period
  The Panic and Agoraphobia Scale (PAS) is self-rating assessing panic disorder and agoraphobia severity with five factor analytic derived subscale scores (panic attacks, anticipatory anxiety, agoraphobic avoidance, health concerns, functional impairment) and a total score indicating the global severity. The questionnaire was specifically developed for monitoring changes during psychotherapy or psychopharmacological treatments. Total score range: 0 to 57. Higher scores indicate worse severity of panic symptomatology.
Change in the severity of anxiety symptomatology (HAM-A= | change from pre-intervention/pre-waiting period (baseline) to immediately after CBT or waiting period
  The Hamilton Anxiety Rating Scale (HAM-A) is a structured clinician rating assessing the severity of anxiety symptomatology. Total score rage: 0 to 56. Higher scores indicate worse severity of anxiety symptomatology.
Change in anxiety sensitivity (ASI) | change from pre-intervention/pre-waiting period (baseline) to immediately after CBT or waiting period
  The Anxiety Sensitivity Index (ASI) is a self-report measure of fear of anxiety-related body symptoms (i.e., anxiety sensitivity). Total score range: 0 to 64. Higher scores indicate worse anxiety sensitivity.

SECONDARY OUTCOMES:
Change in agoraphobic avoidance (MI) | change from pre-intervention/pre-waiting period (baseline) to immediately after CBT or waiting period
  Mobility inventory (MI) is a self-report measure that assess agoraphobic avoidance. Total score range: 1 to 5. Higher scores indicate worse agoraphobic avoidance.
Change in Clinical global impression (CGI) (adapted for panic disorder symptomatology) | change from pre-intervention/pre-waiting period (baseline) to immediately after CBT or waiting period
  Clinical global impression scale (CGI) is a clinician rated global panic disorder severity measure. Total score range: 1 to 7. Higher scores indicate worse global panic disorder severity.
Change in depression symptomatology (BDI) | change from pre-intervention/pre-waiting period (baseline) to immediately after CBT or waiting period
  Beck Depression Inventory (BDI) measures depressive symptomatology (self-report measure). Total score range: 0 to 63. Higher scores indicate worse depressive symptomatology.
Change in Agoraphobic Cognitions (ACQ) | change from pre-intervention/pre-waiting period (baseline) to immediately after CBT or waiting period
  Agoraphobic Cognitions Questionnaire (ACQ) is a self-report measure assessing agoraphobic cognitions. Total score range: 1 to 5. Higher scores indicate worse agoraphobic cognitions.
Change in fear of body symptoms (BSQ) | change from pre-intervention/pre-waiting period (baseline) to immediately after CBT or waiting period
  Self reported fear of body symptoms is measured using the Body Sensation Questionnaire (BSQ). Total score range: 17 to 85. Higher scores indicate worse fear of anxiety sen.

CONTACTS AND LOCATIONS:
Overall Officials: Alfons Hamm, Ph.D., Principal Investigator — Department of Psychology, University of Greifswald
Locations (1):
- University of Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No